CLINICAL TRIAL: NCT06885554
Title: Adjustment Disorders in the US Military: Disease Trajectories and ADNM-20-Mil Validation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USUHS.2024-132; MO240171 (Other Grant/Funding Number: Military Operational Medicine Research Program)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Adjustment Disorders
Keywords: Adjustment Disorders; Military
MeSH Terms: conditions — Adjustment Disorders

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- SANA + Standard of Care (SOC) (Experimental): Participants will be asked to use the SANA device and the Empatica monitoring bracelet for 28 days
  Interventions: Device: SANA
- Standard of Care (SOC) (No Intervention): Participants will be asked to use the Empatica monitoring bracelet for 28 days

INTERVENTIONS:
Device: SANA — SANA is an audio-visual stimulation device found to reduce symptoms commonly found in AjDs. SANA is an eye mask that delivers coordinated pulses of light and sound that facilitate relaxation in the wearer. The device's mechanism of action is neuromodulation through audiovisual stimulation (AVS). When the brain receives a stimulus through the eyes or ears, it emits a responsive electrical charge, called a Cortical Evoked Response (CER). The brain responds by synchronizing to it, a process known as Frequency Following Response (FFR). FFR can be used to trigger each electrical pattern to facilitate a state of relaxation. The Sana device utilizes AVS to induce FFR.
  Arms: SANA + Standard of Care (SOC)

SUMMARY:
Adjustment disorders (AjDs) - a group of mental health diagnosis given following exposure to a stressor that results in preoccupation, failure to adapt, and/or functional impairments - have consistently remained the most common mental health diagnoses in the US military across branches for more than a decade. AjDs can be dangerous and negatively affect military readiness by reducing availability of members and through use of resources to allow evacuations from combat. Diagnosing AjDs can be challenging as it is closely related to other well-defined mental health disorders and assessment and research on AjDs have historically been difficult due to the lack of clarity in the disorder's diagnostic criteria. However, the Adjustment Disorder New Module (ADNM-20) is a recently developed instrument that has shown promise.

In previous work, our team adapted the ADNM-20 to the US military population after finding that there was a need for an AjD-specific diagnostic instrument in this population; this instrument is referred to as the ADNM-20-Mil. The principal focus of this study is the longitudinal psychometric validation of the ADNM-20-mil. However, another goal of the proposed study is to pilot test the audio-visual stimulation device SANA for AjD as pilot testing such a device for AjD is a needed next step. Furthermore, the proposed, longitudinal study provides an ideal platform to test the ADNM-20-Mil's sensitivity to change in the context of this pilot trial to address this critical area of need.

DETAILED DESCRIPTION:
The aim of this trial is to evaluate the sensitivity of the ADNM-20-mil to change via a prospective longitudinal 2-arm repeated measures design to pilot test the feasibility and efficacy of the audio-visual stimulation device SANA. SANA will be used twice daily as an adjunct to standard of care (SOC) within 4-time assessments compared to SOC. Participants will be randomized into a SOC or SOC+Sana group.

Participants in the SOC+SANA arm will be expected to use the SANA device twice daily for 22 minutes per session, with one session just prior to bedtime, from day 1 through day 28 of the T1a period. Both arms of will be expected to wear the Emaptica device 22 hours per day from day 1 through day 28 of the T1a period.

Participants will complete measures at Baseline/T1, 28days/T1a (immediately post-device use), 3months/T2 (2-months post-device use or 3-months post baseline), and 6months/T3 (5-months post device-use or 6-months post baseline).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64
* Serving as active duty in the US Military
* Diagnosed with adjustment disorder (with or without depression and/or anxiety) within the last 3 months
* No other mental health diagnosis (e.g., schizophrenia spectrum and other psychotic disorders, substance use disorder, bipolar and related disorders, TBI)
* No current thoughts of or serious risk of suicide
* Willing and available (e.g., no upcoming deployments or station changes within the next 6 months) to be participate in all study activities if eligible and enrolled
* Any psychotropic drug therapy regimen must be stable (unchanging) for at least 4 weeks prior to enrollment and remain steady throughout the study
* Must have and be willing to use an internet-enabled smartphone or tablet for the study
* Provision of appropriate storage and charging for study equipment in a generally safe and dry condition
* In treatment through the Military Health System for adjustment disorder

Exclusion Criteria:

* Significant medical conditions or other circumstances which would preclude compliance with the protocol, adequate cooperation in the study or obtaining informed consent, or may prevent the patient from safely participating in study.
* Does not meet the eligibility criteria
* Unable to read, speak, or comprehend English
* Unable or unwilling to give informed consent
* No current pregnancy or intention/planned pregnancy during study duration, or lactation
* Study participants of childbearing potential who are unwilling to use an effective method of contraception during the use of SANA device
* History or presence of photo-sensitive epilepsy or other photo-sensitive condition
* History or presence of condition(s) that may affect balance, such as seizure disorders or vertigo
* History or presence of severe and continuous tinnitus
* History or presence of migraine headaches
* Surgery or trauma requiring rehabilitation within the last 12 weeks
* Presence of cancer pain, acute pain following injury or other severe pain that would be anticipated to change during the course of the study
* Vision impairments that affect perception of light, color, or brightness in one or both eyes, and differences in visual perception between eyes
* Deafness in one or both ears, perceived differences in hearing between ears
* Current ear or eye infection, untreated allergies, or acute illness that may affect eyes or hearing (e.g., due to congestion)
* Presence of inflammation or broken skin around the eyes in the area of the mask
* Presence of narcolepsy or untreated sleep apnea. Note: presence of sleep apnea is permitted, so long as patients feel comfortable to use both apnea mask and Sana device in conjunction.
* Participation in any other clinical study in which medication(s) are being delivered or have used an investigational drug or device within the last 30 days.
* Current thoughts of suicide

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Adjustment Disorder-New Module 20 for Military (ADNM-20-Mil) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The ADNM-20-Mil assesses symptoms of AjDs. It consists of two parts: The first part lists a number of stressful life events from which the participant identifies the most distressing event, and the second part lists 20 symptoms that are grouped into six subscales. Each item is rated on a 4-point Likert type scale that rates symptom frequency ranging from 1 (never) to 4 (often) with higher scores indicating worst severity of symptoms. The ADNM-20-mil will be collected via self-report.
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) | Baseline/T1, 3months/T2, 6months/T3
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a structured interview that assesses the severity of PTSD symptoms. The CAPS-5 will be administered to participants via a member of the CAPS-5 study team. This is not a scaled measure as it is a clinical interview.
PTSD Checklist for DSM-5 (PCL-5) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The PCL-5 is a standard 20-item assessment that will be used to assess the presence and severity of PTSD symptoms. Items on the PCL-5 correspond with the DSM-5 criteria for PTSD. Items are rated on a 5-point scale and responses range from 0 (not at all) to 4 (extremely). A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. DSM-5 symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster. The PCL-5 will be collected via self-report.
Adjustment Disorder Diagnosis | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  License healthcare provider diagnosis of adjustment disorder from medical record assessed as the presence or absence of the affiliated ICD-10 or DSM-5 diagnostic code in the medical record. This will be collected retrospectively.

SECONDARY OUTCOMES:
General Well-Being Schedule (GWB) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The GWB is a standard assessment that will be used to measure participants' selfreported positive well-being. The GWB consists of 18 items that are further organized into 6 domains. Out of 18 items, 14 use a 6-point Likert-type scale and represent either intensity or frequency. The four remaining items use a 0-to-10-point rating scale that has opposing adjectives at each end. The total possible scores on the GWB can range from 0 to 110, with higher scores indicating positive well-being. GWB scores can indicate three levels of well-being: score ranges from 0 to 60 indicate "severe distress", score ranges from 61 to 72 indicate "moderate distress", and score ranges from 73 to 110 indicate "positive well-being". The GWB will be collected via self-report.
Depression Anxiety Stress Scales 21 (DASS-21) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The DASS-21 is a standard assessment that will be used to measure participants' selfreported levels of depression, anxiety, and stress. The DASS-21 consists of 21 items and three scales: Depression, Anxiety, and Stress. Each scale has 7 items each rated on a 4-point Likerttype scale ranging from 0 (never) to 3 (almost always) with higher scores indicating greater severity. The DASS-21 will be collected via self-report.
Clinical Global Impression (CGI) | Baseline/T1, 3months/T2, 6months/T3
  The CGI scale is a standard, well-validated measure that provides a clinician's view of the global assessment of how ill their patient is. It consists of 2 items: the CGI-Severity (CGI-S) which measures the severity of the patient's illness on a 7-point rating scale (ranging from normal to very severely ill) and the CGI-Improvement (CGI-I) which measures the patient's overall improvement from baseline also on a 7-point rating scale (ranging from very much worse to very much improved). The higher the scores indicate overall betterment in illness and improvement from baseline. The CGI will be administered to participants via a member of the study team.
Generalized Anxiety Disorder-7 items (GAD-7) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The GAD-7 is a standard assessment of anxiety and will be used to measure anxiety severity and identify participants with a probable actual diagnosis of generalized anxiety disorder. The GAD-7 is a standard clinical measure that is given to MHS patients by their behavioral health provider to complete at every visit. The GAD-7 consists of 7 items with scores that range from 0 to 4 and total score ranging between 0 and 21. The GAD-7 cutoff of >=10 indicates a probable GAD diagnosis. The GAD-7 will be collected retrospectively.
Patient Health Questionnaire-9 items (PHQ-9) | Baseline/T1, 28days/T1a, 3months/T2, 6months/T3
  The PHQ-9 is a standard assessment that will be used to measure depression severity and identify participants with a probable actual diagnosis of major depression. The PHQ-9 is a standard clinical measure that is given to MHS patients by their behavioral health provider to complete at every visit. The PHQ-9 has a cutoff of >=10 for probable depression and its scores can range from 0-27, with higher scores indicating worse depression severity. The PHQ-9 will be collected retrospectively.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Navy Medicine Readiness and Training Command San Diego, San Diego, California
  - Wright Patterson Air Force Base, Wright-Patterson Air Force Base, Ohio
  - Brooke Army Medical Center, Fort Sam Houston, Texas

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT06885554/ICF_001.pdf